CLINICAL TRIAL: NCT00336388
Title: Introduction of Malaria Rapid Diagnostic Tests, Artemisinin-based Combination Therapy, and Malaria Case Management Guidelines at Health Facilities in Kenya: A Cluster Randomized Trial to Evaluate Adherence and Acceptance by Health Care Workers, Impact on Antimalarial Prescription Practices, and Patient Perceptions
Brief Title: Use of Rapid Diagnostic Tests for Malaria Case Management in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); Kenya Division of Malaria Control (Unknown); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDC-NCID-4701
Record Dates: First submitted 2006-06-10; First posted 2006-06-13 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Device: Paracheck Device

SUMMARY:
The purpose of this study is to investigate the impact of rapid diagnostic tests (RDTs) in the context of a newly implemented malaria case management guidelines using artemisinin-based combination therapy on the malaria prescribing practices of health care workers in Kenya.

DETAILED DESCRIPTION:
Malaria causes an estimated 300-500 million infections and over 1 million deaths per year, predominantly in children <5 years old in sub-Saharan Africa. In most parts of malaria endemic sub-Saharan Africa, clinical or presumptive diagnosis, often based on the presence of fever, is the primary means of diagnosing malaria. Clinical diagnosis is sensitive but poorly specific, leading to substantial over-diagnosis. Personnel and supplies to perform microscopic examination of blood smears of persons suspected of having malaria (the current gold standard for diagnosis of malaria) are not available at most health facilities. Over-diagnosis and subsequent over-treatment of patients as a result of clinical diagnosis can lead to increased drug pressure that may facilitate the development of drug resistance in P. falciparum, the malaria parasite responsible for most associated morbidity and mortality in sub-Saharan Africa. This may also increase costs, particularly with the shift from inexpensive antimalarials (such as chloroquine and sulfadoxine-pyrimethamine) to newer, more expensive artemisinin-based combination therapies (ACTs) (such as artemether plus lumefantrine, also known as Coartem®). Over-diagnosis also exposes patients to the unnecessary risk of adverse drug events and, among some patients, leaves the real cause of illness untreated.

Rapid diagnostic tests (RDTs) use immunochromatographic methods to detect antigens derived from malaria parasites in lysed blood. RDTs have generally been reported to achieve field sensitivities and specificities of >90% in the detection of Plasmodium falciparum at densities above 100 parasites/μL blood. RDTs are easy to use and interpret, do not require electricity or special equipment, and can be shipped and stored at ambient conditions.

We hypothesize the use of RDTs should improve malaria diagnosis compared to the use of clinical diagnosis alone. Having access to a test that quickly confirms or excludes the presence of malaria parasites will enable the health care worker (HCW) to determine whether antimalarials are appropriate. If test results are used in this manner, the number of unneeded antimalarial prescriptions should diminish, thus reducing the potential for the development of drug resistance. However, whether and how HCWs will actually use RDT results is unknown. Prior research has demonstrated that results of microscopy are often ignored, and that HCWs often rely on their clinical impressions to diagnose malaria and prescribe treatment.

This study seeks to the describe behaviors and perceptions associated with the use of RDTs for diagnosis of malaria among patients >5 years of age at health facilities in Bondo and Kericho Districts of Kenya, areas of low and high malaria transmission. The specific objectives are:

1. To evaluate the impact of RDTs introduced in the context of newly implemented malaria case management guidelines using ACTs compared to new malaria case management guidelines using ACTs and clinical diagnosis on malaria diagnosis and prescribing practices by HCWs caring for patients >5 years of age.
2. To evaluate HCW performance and adherence to the newly implemented guidelines and use of RDTs.
3. To analyze the costs to a health facility of treating a patient with a fever with two management strategies (RDTs + ACTs compared to clinical diagnosis + ACTs) if treatment guidelines are correctly followed and based on actual HCW adherence to the new guidelines.
4. To evaluate the sensitivity and specificity of RDTs in the hands of HCWs at health facilities in Kenya compared to expert microscopy and compared to RDTs performance in hands of trained study laboratory technicians.
5. To evaluate factors influencing the acceptability of RDTs by HCWs.
6. To evaluate factors influencing the acceptability of RDTs by patients.
7. To evaluate the programmatic implications of RDT introduction.

This trial will generate important public health information regarding the use of RDTs in malaria case management. The study findings will be used to guide provider training, the development of community Information, Education and Communication strategies, and other interventions. These data will be valuable to other countries in sub-Saharan Africa preparing for the introduction of new drug treatment policies and considering methods to improve malaria diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All ill persons >5 years old attending health facilities in Bondo and Kericho Districts, Kenya

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3600
Dates: Start 2006-07; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of malaria diagnosis 6 weeks after the introduction of malaria rapid diagnostic tests

SECONDARY OUTCOMES:
Adherence to malaria case management guidelines by health care workers
Cost effectiveness of malaria case management guidelines using malaria rapid diagnostic tests
Acceptability of malaria rapid diagnostic tests to health care workers
Acceptability of malaria rapid diagnostic tests to patients

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hamel, MD, Principal Investigator — Centers for Disease Control and Prevention; Alexandre Macedo De Oliveira, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Bondo and Kericho District Health Facilities, Kisumu, Nyanza Province, Kenya

REFERENCES:
- [Background] Moody A. Rapid diagnostic tests for malaria parasites. Clin Microbiol Rev. 2002 Jan;15(1):66-78. doi: 10.1128/CMR.15.1.66-78.2002. PMID 11781267